CLINICAL TRIAL: NCT00219245
Title: A 26-Week Open-Label Extension to Protocol No. CENA713BUS11: A 12-Week, Prospective, Double-blind, Placebo-controlled, Multi-center Study Evaluating the Efficacy and Safety of Rivastigmine 3 to 6 mg/Day in Patients With Traumatic Brain Injury (TBI) With Persistent Cognitive Deficits
Brief Title: An Extension Study Evaluating the Efficacy and Safety of Rivastigmine in Patients With Traumatic Brain Injury (TBI) With Persistent Cognitive Deficits
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: CENA713BUS11E1
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Traumatic Brain Injury With Persistent Cognitive Deficits
Keywords: Traumatic brain injury, head trauma, rivastigmine, cognitive deficits
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma; Cognition Disorders | interventions — Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine

SUMMARY:
Patients who completed the 12-week double blind protocol may enter this 26-week, open-label extension. This extension will give patients who complete the study an opportunity to receive treatment with open-label rivastigmine 3-12 mg/day and further evaluation for the cognitive deficits related to traumatic brain injury. This extension will enable further evaluation of patients, as well as analyses to be conducted examining response to treatments in the original drug and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Have a deficit in the areas of attention and/or memory.
* Have current cognitive deficits which were present from the time of the injury, are persistent, and are deemed to be the result of the brain injury;
* Be at least 12 months post brain injury;

Exclusion Criteria:

* A history of a major brain surgery;
* A penetrating brain injury (e.g., gun shot wound);
* A current diagnosis of epilepsy;
* Had more than one seizure in the past year (patients who have had a single seizure within a year post-injury will be considered on a case by case basis);
* Previous exposure to rivastigmine.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2002-11; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Improvement in cognitive functioning in the areas of attention or verbal memory from baseline to week 26
Safety and tolerability of 26 week's of treatment with rivastigmine in patients with traumatic brain injury with persistent cognitive impairment

SECONDARY OUTCOMES:
Changes in cognitive functioning from baseline to week 26
Changes in behavior from baseline to week 26
Changes in depression from baseline to week 26
Changes in quality of life from baseline to week 26
Changes in overall functioning from baseline to week 26

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Sponsor GmbH